CLINICAL TRIAL: NCT06193759
Title: Immunotherapy for Malignant Pediatric Brain Tumors Employing Adoptive Cellular Therapy (IMPACT)
Acronym: IMPACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Medulloblastoma, Childhood; Atypical Teratoid/Rhabdoid Tumor of CNS; Embryonal Tumor With Multilayered Rosettes; Pineoblastoma; Embryonal Tumor of CNS
MeSH Terms: conditions — Medulloblastoma; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Pinealoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Embryonal brain tumors (Experimental): These patients are young children (<5 years of age) with newly diagnosed high-risk embryonal CNS malignancies and are expected to have a modest male predominance reflecting the sex-based incidence of pediatric brain tumors. Patients will have a Lansky performance status of ≥60.
  Interventions: Biological: Multi-tumor antigen specific cytotoxic T lymphocytes (TSA-T) directed against proteogenomically determined personalized tumor-specific antigens (TSA)

INTERVENTIONS:
Biological: Multi-tumor antigen specific cytotoxic T lymphocytes (TSA-T) directed against proteogenomically determined personalized tumor-specific antigens (TSA) — Young patients with embryonal central nervous system (CNS) malignancies typically are unable to receive irradiation due to significant adverse effects and are treated with intensive chemotherapy followed by autologous stem cell rescue; however, despite intensive therapy, many of these patients relapse. In this study, individualized TSA-T cells will be generated against proteogenomically determined tumor-specific antigens after standard of care treatment in children less than 5 years of age with embryonal brain tumors.

SUMMARY:
This is an open-label phase 1 safety and feasibility study that will employ multi-tumor antigen specific cytotoxic T lymphocytes (TSA-T) directed against proteogenomically determined personalized tumor-specific antigens (TSA) derived from a patient's primary brain tumor tissues. Young patients with embryonal central nervous system (CNS) malignancies typically are unable to receive irradiation due to significant adverse effects and are treated with intensive chemotherapy followed by autologous stem cell rescue; however, despite intensive therapy, many of these patients relapse. In this study, individualized TSA-T cells will be generated against proteogenomically determined tumor-specific antigens after standard of care treatment in children less than 5 years of age with embryonal brain tumors. Correlative biological studies will measure clinical anti-tumor, immunological and biomarker effects.

DETAILED DESCRIPTION:
This study will be conducted at Children's National Hospital (CNH) in Washington, DC. TSA-T products will be manufactured at the cell therapy Good Manufacturing Practice (GMP) facility at CNH. Patients enrolled in the study will receive their infusions at CNH.

This is a phase 1 study treating children with embryonal brain tumors after definitive resection. Residual tumor may be present at the primary site or metastatic deposits but is not required.

Patients will be treated with standard of care therapy as required, which may include up to 3 induction chemotherapy cycles (vincristine, cyclophosphamide, cisplatin, etoposide with or without methotrexate) and up to 3 consolidation cycles (carboplatin and thiotepa, each followed by an infusion of autologous peripheral blood stem cells (PBSCs)). Please note: Methotrexate will be part of the induction chemotherapy as per treating physician's discretion.

The first TSA-T dose will be infused via a Codman Holter Rickham reservoir and catheter (intraventricular access device) on day 0, which will ideally be within 10 days following the patient's blood count recovery (ANC>1000, ALC>500) after the final consolidation cycle. Patients will receive the TSA-T product as per the table below until the recommended phase 2 dose (RP2D) is reached.

Three patients will be enrolled at dose level 1 (2.5x107 cell) and monitored for at least 42 days during the safety monitoring period. If 2 DLTs are observed, the dose will be de-escalated to dose level -1 (1x107 cells). If no DLT is observed, 3 more patients will be enrolled at dose level 2 (5x107 cells). If 1 DLT is observed, an additional 3 patients will be enrolled at dose level 1 (2.5x107 cell) to complete the 42-day safety monitoring period. After these first 6 patients, an interim analysis to evaluate adverse events (AE) will occur. If there are ≤1 DLT in these first 6 patients and no other serious safety concerns, the remainder of the planned enrollment of 12 patients will be enrolled at dose level 2 (5x107 cells). If >1 DLT is observed in the first 6 patients, the dose will be reduced to 1x107 cells, and another 3 patients will be enrolled and monitored for the 42-day safety monitoring period. If no further DLTs are encountered, the remainder of the planned enrollment of 12 will be enrolled at 1x107 cells. If any DLTs are observed at 1x107 cells, enrollment will be suspended, and the Data Review Committee (DRC) will meet to determine the feasibility of a further dose reduction. For the 3 patients treated at dose level 2 (5x107 cells), similarly if 1 DLT is observed, additional 3 patients will be enrolled at this dose level. If >1 DLT is observed out of the 6 patients, the dose will be de-escalated to dose level 1, and the remainder of the patients will be enrolled at 2.5x107 cells. Each patient will receive at least one TSA-T infusion and may receive a maximum of 8 total infusions if sufficient TSA-T cells are available. For any infusion following the first infusion, if a patient's TSA-T supply is insufficient to meet the dose at the enrollment dose level, the final infusion may be administered at a lower dose level at the treating physician's discretion. The first and second infusions will be administered at least 42 days apart and additional infusions will be spaced at least 28 days apart. If patients have a response of stable disease or better by iRANO criteria at the evaluation after the second infusion OR if they have clinical stability and a clinical assessment of possible pseudoprogression on MRI despite the appearance of radiographic progression (see below), they are eligible to receive up to 6 additional infusions of TSA-T at a minimum of 28-day intervals as long as TSA-T cells are available. Each additional infusion will be the same as the enrollment dose level (i.e., no subsequent dose escalation).

Prior to the first infusion, if a patient's TSA-T supply is insufficient for the dose level that the patient is assigned to, the patient may receive TSA-Ts at a lower dose with a minimum of 1x107 cells. These patients will not count towards the overall safety objective and will be replaced for that objective, although they will count towards the feasibility objective of identifying and producing adequate TSA-T products. If patients who are clinically stable are deemed to have possible pseudoprogression, then these patients may still be eligible for infusion if serial imaging and clinical assessments demonstrate stability most consistent with pseudoprogression. In these patients, disease assessment after the imaging that first raises the concern for pseudoprogression (potential progressive disease versus pseudoprogression) must be at least stable compared with the initial scan demonstrating enlarging tumor size.

ELIGIBILITY:
Inclusion Criteria:

RECIPIENT PROCUREMENT (BLOOD COLLECTION FOR TSA-T MANUFACTURING) INCLUSION CRITERIA

* New diagnosis of CNS embryonal tumors: medulloblastoma, embryonal tumor with multilayered rosettes (ETMR), pineoblastoma, atypical teratoid/rhabdoid tumor, and embryonal tumor, not otherwise specified (NOS).
* <5 years of age at enrollment.
* Lansky score of ≥60% (see appendix B).
* Organ function:

ANC ≥750/µL. Absolute lymphocyte count (ALC) >500/μL. Platelets ≥75K. Bilirubin ≤3xULN. Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) <5x upper limit of normal (ULN). Serum creatinine ≤1.0mg/dL or 1.5x ULN for age (whichever is higher). Pulse oximetry >90% on room air.

* Parent(s)/guardian(s) capable of providing informed consent.
* Availability of sufficient pre-trial fresh frozen tumor tissue (approximately 50 mg).
* Patient deemed to be of sufficient size to undergo PBMC pheresis for TSA-T generation and PBSC rescue.
* Patient is a surgical candidate for placement of Rickham reservoir in the opinion of a physician.

RECIPIENT INCLUSION CRITERIA FOR INITIAL TSA-T ADMINISTRATION AND FOR ADDITIONAL INFUSIONS

* Lansky score of ≥60%.
* Organ function:

Bilirubin ≤3x ULN. AST/ALT ≤5x ULN. Serum creatinine ≤1.0mg/dL or 1.5x ULN for age (whichever is higher). Pulse oximetry >90% on room air.

- Neurologic status: Patient must have a stable neurologic exam for 2 weeks, on a stable or decreasing dose of steroids, prior to administration of the first dose of TSA-T cells, and stability for 1 week prior to all subsequent infusions. The exams demonstrating stability must be performed by the study team, although these may occur via telemedicine if necessary. Patient must agree to a brief (<72 hours) course of steroids

Exclusion Criteria:

PROCUREMENT EXCLUSION CRITERIA

* Patients with uncontrolled infections.
* Patients with known HIV infection.
* Prior immunotherapy with an investigational agent within the last 28 days prior to procurement.
* Patients with medulloblastoma of the SHH subtype.
* Patients who have overly bulky tumors on imaging are ineligible. These include the following:

Tumor with any evidence of herniation or significant midline shift. Tumor with a significant brainstem component. Patients who are deemed to have overly bulky tumor by the principal investigator (PI) of the study.

RECIPIENT EXCLUSION CRITERIA FOR INITIAL AND SUBSEQUENT TSA-T INFUSIONS

* Patients with uncontrolled infections.
* Patients who have overly bulky tumors on imaging are ineligible. These include the following:

Tumor with any evidence of herniation or significant midline shift. Tumor with a significant brainstem component. Patients who are deemed to have overly bulky tumor by the PI of the study.

* Patients who received ATG, Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of TSA-T infusion.
* Patients receiving dexamethasone at a dose of >0.05mg/kg. All patients who qualify based on the above inclusion and exclusion criteria will be eligible for participation in this study.

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2030-12-29 (Estimated); Study Completion 2032-12-29 (Estimated)

PRIMARY OUTCOMES:
Grade ≥3 infusion-related adverse event | 42 days of the first TSA-T infusion
  Number of patients with Grade ≥3 infusion-related adverse event (per CTCAE version 5) occurring within 42 days of the first TSA-T infusion.
Grade ≥4 non-hematologic adverse event | 42 days of the first TSA-T infusion
  Number of patients with Grade ≥4 non-hematologic adverse event (per CTCAE version 5) occurring within 42 days of the first TSA-T infusion that is not due to the patient's underlying malignancy or chemotherapy related co-morbidities. Toxicities that do not resolve with bone marrow recovery (defined as an absolute neutrophil count (ANC) >1000) may be possibly related to the TSA-T therapy.
Grade ≥3 pneumonitis, uveitis | 42 days of the first TSA-T infusion
  umber of patients with grade ≥3 pneumonitis, uveitis (per CTCAE version 5)
Grade ≥3 toxicities that are attributed to TSA-T | 42 days of the first TSA-T infusion
  Number of patients with grade ≥3 toxicities (CTCAE version 5) that are attributed to TSA-T. (Toxicities that do not resolve with bone marrow recovery (defined as an ANC >1000) may be possibly related to the TSA-T therapy.).
Any unexpected toxicity of grade ≥3 attributed to the infusion of TSA-T | 42 days of the first TSA-T infusion
  Number of patients with any unexpected toxicity of grade ≥3 (per CTCAE version 5) attributed to the infusion of TSA-T

SECONDARY OUTCOMES:
TSA-T responses | 1 Year
  Determine the number of patients who respond to TSA-T
Progression free survival | 5 years
  The interval of time between the date of protocol treatment initiation and the earliest date of documentation of progressive disease, or second malignancy or death (for any reason) for patients who fail, or to date of last contact or initiation of other therapy for patients who remain at risk of failure.
Overall survival | 5 years
  Overall survival post last TSA-T infusion

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Hwang, MD, Principal Investigator — Children's National Research Institute; Brian Rood, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No